CLINICAL TRIAL: NCT03609710
Title: The Effect of Combined Application of Left Colic Artery Preservation, Anastomotic Reinforcing Sutures and Transanal Tube Placement in Robotic Low Anterior Resection for Rectal Cancer to Prevent Anastomic Leak：A Prospective, Single-center, Randomized Control Trial Study
Brief Title: Application of Left Colic Artery Preservation, Anastomotic Reinforcing Sutures and Transanal Tube in Robotic Low Anterior Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Prof., Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSTLAR
Record Dates: First submitted 2018-07-23; First posted 2018-08-01 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-01

CONDITIONS: Rectal Cancer
Keywords: Low rectal cancer; Robotic surgery; Anastomotic leak
MeSH Terms: conditions — Rectal Neoplasms; Anastomotic Leak | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PSTLAR (Experimental): Combined application of left colic artery preservation, anastomotic reinforcing sutures and postoperative transanal tube placement in robotic low anterior resection for rectal cancer
  Interventions: Device: Transanal tube placement; Procedure: Left colic artery preservation; Procedure: Anastomotic reinforcing sutures; Device: Robotic surgery
- NORLAR (Active Comparator): Traditional robotic low anterior resection for rectal cancer without left colic artery preservation, anastomotic reinforcing sutures or postoperative transanal tube placement
  Interventions: Device: Robotic surgery

INTERVENTIONS:
Device: Transanal tube placement — Transanual tube placement after anastomosis in low anterior resection for rectal cancer.
  Arms: PSTLAR
Procedure: Left colic artery preservation — Left colic artery preservation during operation for lower rectal cancer
  Arms: PSTLAR
Procedure: Anastomotic reinforcing sutures — Anastomotic reinforcing sutures during operation for lower rectal cancer
  Arms: PSTLAR
Device: Robotic surgery — Robotic low anterior resection for rectal cancer

SUMMARY:
The purpose of this study is to evaluate the results of combined application of left colic artery preservation, anastomotic reinforcing sutures and postoperative transanal tube placement in robotic Low Anterior Resection for Rectal Cancer.

DETAILED DESCRIPTION:
Combined application of left colic artery preservation, anastomotic reinforcing sutures and postoperative transanal tube placement in robotic low anterior resection for rectal cancer

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of low rectal cancer; Low rectal cancer was defined by the presence of the inferior pole of the tumor below the peritoneal reflection (in 11 cm from the anal margin)
* Primary tumor has undergone histologically comfirmed rectal adenocarcinoma
* Together with clinical or radiological evidence of Stage II (T3-4, N0, M0) or Stage III (T1-4, N1-2, M0) disease (according to the 2016 revision of the International Union Against Cancer primary tumor, regional nodes, metastasis (TNM) staging system)
* Performance status (ECOG) 0~1
* Adequate hematological function: Neutrophils≥1.5 x109/l and platelet count≥100 x109/l; hemoglobin (Hb) ≥9g/dl (within 1 week prior to randomization)
* Adequate hepatic and renal function: Serum bilirubin≤1.5 x upper limit of normal (ULN), alkaline phosphatase ≤5x ULN, and serum transaminase (either primary tumor, regional nodes, metastasis (AST) or ALT) ≤ 5 x ULN(within 1 week prior to randomization);
* Written informed consent for participation in the trial.

Exclusion Criteria:

* Body mass index (BMI) more than 30 kg/m2
* Serious pre-operative comorbidity, including cardiovascular disease (coronary arteriosclerosis, arrhythmia, heart failure), pulmonary dysfunction (lung emphysema, obstructive lung disease), liver insufficiency (Child-Pugh B or C), renal insufficiency (serum creatinine >2.0 mg/dl), and arterial circulation disturbance (occlusion of arterial vessels of limb in patient's history
* History of accepting abdominal surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-05-30 (Estimated)

PRIMARY OUTCOMES:
Anastomotic leak rate | 30 days post operatively
  Anastomotic leak is a common and serious complication after low anterior, resection, and often leads to re-operation.

SECONDARY OUTCOMES:
Reoperation rate after anastomotic leak | 30 days post operatively
  Anastomotic leak is a common and serious complication after low anterior, resection, and often leads to excrement peritonitis, and re-operation as colostomy

CONTACTS AND LOCATIONS:
Locations (1):
- Jianmin Xu, Shanghai, Shanghai Municipality, China